CLINICAL TRIAL: NCT04383860
Title: Choice of Sutures in Orbital Implants in Retinoblastoma Patients
Brief Title: Sutures in Orbital Implants in Retinoblastoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Surgery--Complications; Retinoblastoma Bilateral
Keywords: Retinoblastoma; suture; complications
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-0 suture (Experimental): 5-0 suture administration during surgery
  Interventions: Procedure: 5-0 suture
- 4-0 suture (Active Comparator): 4-0 suture administration during surgery
  Interventions: Procedure: 4-0 suture

INTERVENTIONS:
Procedure: 5-0 suture — 5-0 suture administration during surgery
  Other Names: 5-0 suture administration
  Arms: 5-0 suture
Procedure: 4-0 suture — 4-0 suture administration during surgery
  Other Names: 4-0 suture administration
  Arms: 4-0 suture

SUMMARY:
The purpose of this study is to evaluate different sutures for orbital implants in retinoblastoma patients.

DETAILED DESCRIPTION:
To evaluate the effectiveness and complications of 4-0 and 5-0 sutures for orbital implants in retinoblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as retinoblastoma
* enucleation and orbital implantation in the same surgery

Exclusion Criteria:

* death during follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of participants with complications | 2 year after surgery
  complications, such as orbital implant exposure in the follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No